CLINICAL TRIAL: NCT07126782
Title: Clinical Study on the Efficacy and Safety of Allogeneic γδ T Cells in the Treatment of Patients With MRD-positive Acute Myeloid Leukemia (AML) After Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT)
Brief Title: The Efficacy and Safety Assessment of Allogeneic γδ T Cells in Patients With MRD-positive AML After Allo-HSCT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025056
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-06

CONDITIONS: AML (Acute Myelogenous Leukemia); AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic γδ T cell immunotherapy (Experimental): Patients will receive at least 4 cycles of in vitro extended allogeneic γδ T cell therapy, twice a week.
  Interventions: Biological: Ex-vivo expanded allogeneic γδ T cells

INTERVENTIONS:
Biological: Ex-vivo expanded allogeneic γδ T cells — Cells will be extracted from a healthy donor by apheresis, followed by ex-vivo expansion and activation. The ex-vivo expanded γδ T cells from donors will be adoptively transfused.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of allogeneic γδ T cells in patients with MRD-positive AML after allo-HSCT.

DETAILED DESCRIPTION:
This is a single-center, randomized, open label phase I clinical trial to evaluate the efficacy and safety of ex-vivo expanded allogeneic γδ T cells in patients with MRD-positive AML after allo-HSCT. The infusion doses of γδ T cells were 2E8 cells/kg and 4E8 cells/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should sign informed consent form voluntarily before the trail and comply with the requirements of this study.
2. Age≥18 years old, gender unlimited.
3. All the subjects met the 2016 WHO classification and were diagnosed with AML via MICM (Morphology,Immunophenotyping, Cytogenetics, and Molecular genetics).
4. AML patients receiving allo-HSCT.
5. Subjects classified into the favorable -to-intermediate risk group according to the 2022 European Leukemia Net (ELN) risk stratification guidelines.
6. All subjects were detected positive for MRD, and MRD was positive by flow cytometry (MFC) or/and positive for fusion genes/gene mutations by RQ-PCR.
7. ECOG performance status score: 0-2.
8. Inactive GVHD (acute GVHD grade II-IV or moderate to severe chronic GVHD).
9. Adequate bone marrow reserve, defined as: absolute neutrophil count (ANC) > 0.5E9/L and platelet count ≥20E9/L.
10. Adequate organ function as per protocol.
11. Male and female patients of reproductive potential must agree to use birth control during the study and for at least 28 days post study.

Exclusion Criteria:

1. Post-transplant relapse or extramedullary disease: AML patients post-allo-HSCT with ≥5% blasts in peripheral blood or bone marrow (excluding causes such as bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemia infiltration.
2. Active GVHD: Subjects with active GVHD within 30 days before screening.
3. Active infections: HBV, HCV, HIV, syphilis (TP), active CMV, or EBV infection.
4. Neurological disorders: active autoimmune or inflammatory neurological diseases, clinically significant active cerebrovascular disease.
5. Unstable systemic diseases, including: unstable angina, cerebrovascular accident or transient ischemic attack (within 6 months before screening), myocardial infarction (within 6 months before screening), NYHA Class III/IV heart failure, refractory hypertension (defined as failure to control blood pressure despite lifestyle modifications and treatment with ≥4 antihypertensive drugs, including diuretics, for >1 month), clinically significant arrhythmias requiring medication, severe hepatic, renal, or metabolic disorders.
6. Major surgery: Subjects who underwent major surgery within 4 weeks before screening, as deemed ineligible by the investigator.
7. Concurrent non-hematologic malignancies.
8. Cardiac abnormalities, meeting any of the following: Left ventricular ejection fraction (LVEF) ≤45%. NYHA Class III/IV congestive heart failure. QTc interval >480 msec. Other cardiac conditions considered unsuitable by the investigator.
9. History of epilepsy or other active CNS disorders.
10. Uncontrolled infections: active systemic infections requiring treatment (e.g., sepsis, bacteremia, fungemia, tuberculosis, opportunistic infections).
11. Recent participation in other interventional trials: Subjects who participated in another interventional clinical study within 30 days prior to enrollment.
12. Other conditions: Any other circumstances deemed by the investigator to compromise subject safety or trial integrity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2028-07-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 4weeks
  Defined as the MRD-negative complete remission rate (CRMRD- rate) at 4 weeks, representing the proportion of subjects achieving MRD negativity after 4 weeks of treatment.

SECONDARY OUTCOMES:
MRD-negative rate at 2 weeks (CRMRD- rate) | 2weeks
  Proportion of subjects achieving MRD negativity after 2 weeks of treatment.
Duration of Response (DOR) | 4weeks
  Time from the first documented MRD-negative complete remission (CRMRD-) to the first occurrence of disease progression or death from any cause. For subjects without confirmed progression or death, DOR will be censored at the last evaluable assessment.
2-Year Overall Survival (OS) | 2 years
  Proportion of subjects who remain alive at 2 years from the first dose of study treatment.
Safety observation | Baseline to 2 years
  Incidence of Grade ≥3 adverse events (AEs) Incidence of GVHD Non-relapse mortality (NRM)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No